CLINICAL TRIAL: NCT06706479
Title: The Effects of High-definition Transcranial Direct Current Stimulation on Balance Control in Older Adults With Chronic Low Back Pain: a Randomized Controlled Trial
Brief Title: The Effects of High-definition Transcranial Direct Current Stimulation on Balance Control in Older Adults With Chronic Low Back Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Arnold Wong Yu Lok, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20240416001
Record Dates: First submitted 2024-08-26; First posted 2024-11-26 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The allocation of the participants will be sealed in an envelope, blinding the subjects and assessors, and a third person (intervention implementer) will perform the blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active stimulation (Experimental): For the active stimulation, the current will be ramped up from 0 to 2 mA over the initial 30-s period and then maintain the current of 2 mA for 20 minutes, following by a 30-s ramp-down period.
  Interventions: Device: high-definition transcranial direct current stimulation
- Sham stimulation (Experimental): The participants will receive the same intervention procedures, but the intervention will have no therapeutic effect. Specifically, for the sham stimulation, participants will only experience 30-s ramp-up and 30-s ramp-down periods at both the commencement and end of the stimulation.
  Interventions: Device: high-definition transcranial direct current stimulation

INTERVENTIONS:
Device: high-definition transcranial direct current stimulation — High-definition transcranial direct current stimulation is a novel non-invasive brain stimulation technique based on the principle that when weak intensity electric currents are targeted on specific areas of the scalp, they cause underlying cortical stimulation. The anode increases cortical excitability, while cathode decreases cortical excitability.

SUMMARY:
The goal of this clinical trial is to investigate the effects and mechanisms of high-definition transcranial direct current stimulation over left dorsolateral prefrontal cortex on chronic low back pain and balance in older adults. The main questions it aims to answer are:

Primary hypothesis 1: Active stimulation would have greater improvement in pain and balance, reduced left dorsolateral prefrontal cortex activation than sham stimulation.

Primary hypothesis 2: Active stimulation would have enhanced functional connectivity than sham stimulation.

Primary hypothesis 3: The balance improvement would be related to reduced pain, decreased left dorsolateral prefrontal cortex activation, enhanced functional connectivity, attention, and/or executive function.

Participants will be randomly received a single-session of high-definition transcranial direct current stimulation (active or sham stimulation). Before and immediately after the intervention, balance (semi-tandem stance and timed up-and-go test (TUG)) and cognitive (attention and executive function) tests will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-85 years;
* With non-specific chronic low back pain that has no definitive diagnosis but lasted for at least 3 months, typically occurs in the area between the lower rib margins and the buttock creases;
* With an average pain intensity over the last week to be ≥ 3 on an 11-point numerical rating scale (NRS) anchored with "no pain" at zero and "worst pain imaginable" at 10;
* Have normal cognitive function (Hong Kong Montreal Cognitive Assessment ≥ 22);
* Who agree to sign an informed consent form.

Exclusion Criteria:

* Inability to ambulate without assistance from another person or tools (e.g., canes or walkers);
* Having specific causes of low back pain (e.g., spinal stenosis, lumbar disc herniation, spondylolisthesis, recent vertebral fracture, spinal infection);
* Having other acute or overt musculoskeletal conditions in other parts of the body (e.g., fractures, severe pain, multiple joint pain (e.g., knee pain));
* History of lumbar or lower extremity surgery;
* Receiving LBP treatment within the past one month or at present;
* Have never received non-invasive brain stimulation (e.g., transcranial direct current stimulation, repetitive transcranial magnetic stimulation, and transcranial alternating current stimulation) before.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Current back-pain intensity | Before and immediately after the intervention.
  The current back-pain intensity will be assessed with the 11-point numerical rating scale anchored with "no pain" at zero and "worst pain imaginable" at 10.

SECONDARY OUTCOMES:
Resting-state blood oxygen concentration | Before and immediately after the intervention.
  Resting-state blood oxygen concentration (indicated by Oxyhemoglobin concentration (μmol)) will be measured using the portable fNIRS imaging system (NIRSport 2, NIRx Medical Technologies LLC, Glen Head, NY, USA). We will instruct participants to sit still and comfortably with their eyes open, lean against the back rest, and look at a fixation cross one meter in front of them for 5 minutes.
Arithmetic performance | Before and immediately after the intervention.
  Participants will be required to perform the cognitive task in the seated postition (3 x 30s). The cognitive task is serial subtraction from a random three-digit number (200-999) by 7s audibly. The number of correct and incorrect answers will be recorded.
Postural sway | Before and immediately after the intervention.
  Postural sway will be assessed by APDM® Mobility Lab (APDM, Inc., Portland, OR, USA) in the following tests in a random order: (1) semi-tandem stance on firm surfaces without cognitive task (3 x 30s), (2) semi-tandem stance on firm surfaces with cognitive task (3 x 30s), (3) semi-tandem stance on foam surfaces without cognitive task (3 x 30s), (4) semi-tandem stance on foam surfaces with cognitive task (3 x 30s). The cognitive task is serial subtraction from a random three-digit number (200-999) by 7s audibly. No instructions are given regarding task prioritization. During the standing tests, cortical activation will be measured using the NIRSport 2 system with its control box placed in a backpack worn by participants.
Timed up-and-go test (TUG) | Before and immediately after the intervention.
  TUG will be performed in random order in the following tests: (1) TUG without a cognitive task (3 trials) and (2) TUG with a cognitive task (3 trials). The cognitive task involves serial subtraction from a random three-digit number (ranging from 200 to 999) by subtracting 7s audibly. No specific instructions are provided regarding task prioritization. The time (in seconds) taken to complete the TUG, along with the number of correct and incorrect answers, will be recorded for statistical analysis.
Attention | Before and immediately after the intervention.
  Attention will be assessed using the Trail Making Test - A (TMT-A). TMT-A involves connecting a series of 25 square and circle encircled numbers in ascending order, without lifting the pen from the paper. Errors will be corrected immediately and re-establish the sequence. The time (in seconds) to complete the TMT-A will be recorded for statistical analysis.
Executive function | Before and immediately after the intervention.
  Executive function will be assessed using TMT-A and the Trail Making Test - B (TMT-B). TMT-A involves connecting a series of 25 square and circle encircled numbers in ascending order, without lifting the pen from the paper. In TMT-B, the numbers from 1 to 25 are twice presented in square and circle shapes ("1" is only presented once). Participants are instructed to connect the numbers in ascending order, alternating between the squares and circles. Errors will be corrected immediately and re-establish the sequence. The time to complete the TMT-A and TMT-B will be recorded. Executive function will be indicated by the difference in TMT-A and TMT-B (TMT-B minus TMT-A in seconds).
Side or adverse effects | During and 1 hour after the intervention.
  Any side or adverse effects (e.g., itching, tingling and burning sensations under electrodes) related to the interventions will be monitored in all participants.
Blinding efficacy | Immediately after the intervention.
  A blinding efficacy questionnaire will be completed after intervention. If the participant believes that they receive active or sham stimulation, they will be asked to state their confidence in this belief on a scale of 1 (not confident) to 3 (very confident).

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No